CLINICAL TRIAL: NCT01385761
Title: A Prospective, Randomized Non- Crossover Investigation of the LMA Unique TM and the Self Pressurized Air-Q TM Intubating Laryngeal Airway in Children
Brief Title: LMA Unique TM & the Self Pressurized Air-Q TM Intubating Laryngeal Airway in Children
Status: Completed | Type: Observational
Sponsor: Ann & Robert H Lurie Children's Hospital of Chicago (Other)
Responsible Party: Principal Investigator, Narasimhan Jagannathan, primary investigator, Ann & Robert H Lurie Children's Hospital of Chicago
Other Study IDs: IRB#2011-14642
Record Dates: First submitted 2011-06-28; First posted 2011-06-30 (Estimated); Last update posted 2012-03-13 (Estimated); Status verified 2012-03

CONDITIONS: Children
Keywords: Supraglottic airway devices
MeSH Terms: interventions — Laryngeal Masks

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Laryngeal Mask airway (LMA): children weighing 20 to 30 kg
  Interventions: Device: Laryngeal Mask Airway
- Intubating Laryngeal Airway (ILA-SP): Children weighing 20-30 kg
  Interventions: Device: air-QTM Intubating Laryngeal Airway

INTERVENTIONS:
Device: Laryngeal Mask Airway — Each child will be randomized to either receiving the LMA or air-Q ILA-SP as their supraglottic airway device for primary airway maintenance.
  Other Names: Laryngeal Mask AirwayTM (Laryngeal Mask Airway North America; San Diego, CA USA)
  Groups: Laryngeal Mask airway (LMA)
Device: air-QTM Intubating Laryngeal Airway — Each child will be randomized to either receiving the LMA or air-Q ILA-SP as their supraglottic airway device for primary airway maintenance.
  Other Names: air-QTM Intubating Laryngeal Airway Mercury Medical;Clearwater, Fl USA
  Groups: Intubating Laryngeal Airway (ILA-SP)

SUMMARY:
The purpose of this study is to compare the clinical efficacy of the air-Q ILA-SP with the current standard of care, the LMA Unique in anesthetized non-paralyzed pediatric patients.

DETAILED DESCRIPTION:
The goal for this randomized, non-crossover investigation is to compare a disposable version of the standard LMA, LMA Unique TM,with the air-Q ILA-SP in pediatric patients. Oropharyngeal leak pressure is commonly used as an indicator of airway seal adequacy. Similarly, flexible fiberoptic bronchoscope examination is often employed to assess proper placement of airway devices. We hypothesize that airway leak pressures with the ILA-SP will be superior to the LMA upon initial device placement, and ten minutes after device placement. Airway leak pressures will be measured by recording the circuit pressure at which equilibrium is reached. Ease of placement, fiberoptic grade of laryngeal view, and complications (airway related, gastric insufflation, trauma) will also be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Children undergoing general anesthesia using a supraglottic airway device
* 3 to 9 years of age
* 20 to 30 kilograms in weight

Exclusion Criteria:

* History of a difficult airway
* Active gastrointestinal reflux
* Active upper respiratory tract infection

Ages: 3 Years to 9 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Children weighing 20 to 30 kg undergoing surgery requiring a supraglottic airway device
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2011-06; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Oropharyngeal leak pressure | 2 months

CONTACTS AND LOCATIONS:
Overall Officials: Narasimhan Jagannathan, MD, Principal Investigator — Childrens Memorial Hospital
Locations (1):
- Childrens Memorial Hospital, Chicago, Illinois, United States

REFERENCES:
- [Background] Jagannathan N, Sohn LE, Mankoo R, Langen KE, Roth AG, Hall SC. Prospective evaluation of the self-pressurized air-Q intubating laryngeal airway in children. Paediatr Anaesth. 2011 Jun;21(6):673-80. doi: 10.1111/j.1460-9592.2011.03576.x. PMID 21518103
- [Background] Shimbori H, Ono K, Miwa T, Morimura N, Noguchi M, Hiroki K. Comparison of the LMA-ProSeal and LMA-Classic in children. Br J Anaesth. 2004 Oct;93(4):528-31. doi: 10.1093/bja/aeh238. Epub 2004 Aug 6. PMID 15298876
- [Background] White MC, Cook TM, Stoddart PA. A critique of elective pediatric supraglottic airway devices. Paediatr Anaesth. 2009 Jul;19 Suppl 1:55-65. doi: 10.1111/j.1460-9592.2009.02997.x. PMID 19572845